CLINICAL TRIAL: NCT03554785
Title: Comparative Effectiveness Research to Improve the Health of Sexual and Gender Minority Patients Through Cultural Competence and Skill Training of Community Health Center Providers and Non-clinical Staff
Acronym: PCORI-SOGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenway Community Health (Other)
Collaborators: OCHIN, Inc. (Other); AllianceChicago (Other); Association of Asian Pacific Community Health Organizations (Unknown); Beaufort Jasper Hampton Comprehensive Health Services (Unknown); Kaiser Permanente (Other); Patient-Centered Outcomes Research Institute (Other); Piedmont Healthcare (Other); Howard Brown Health Center (Other); Heartland Alliance (Other); Near North Health Service Corporation (Unknown); Legacy Health System (Other); Campus Health Center - Wayne State University (Nursing Practice Corporation) (Unknown); Eureka Community Health & Wellness Center (Unknown); Winding Waters Clinic (Unknown); CHARLES B WANG COMMUNITY HEALTH CENTER (Unknown); Waimanalo Health Center (Unknown)
Responsible Party: Principal Investigator, Kenneth H. Mayer, MD, Co-Chair and Medical Research Director, Fenway Community Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 6271
Record Dates: First submitted 2018-05-14; First posted 2018-06-13 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: LGBT Health; Cultural Competency; Education; Sexual Orientation; Gender Identity
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control/Usual Care (No Intervention): * Readiness Assessment (web survey for CHC leadership and providers)
  * Patient web surveys (10 total per site; 5 SGM and 5 cisgendered)
  * Option to view 60 minute online webinar "Do Ask, Do Tell: Collecting Data on Sexual Orientation and Gender Identity at Health Centers"
- Intervention (Active Comparator): * Readiness Assessment (web survey for CHC leadership and providers)
  * Patient web surveys (10 total per site; 5 SGM and 5 cisgendered)
  * CHC staff leadership key informant interviews (up to 5 at each site)
  * Tailored Educational Clinician and Non-clinician staff training intervention and technical assistance follow-up
  Interventions: Behavioral: Clinician and Non-clinician staff training

INTERVENTIONS:
Behavioral: Clinician and Non-clinician staff training — An optimized training program for non-clinical staff, clinicians and administrators developed by TFI's National LGBT Health Education Center that will include content-specific webinars and "Office Hours" for specific CHC consultations to optimize the provision of SGM health services at each CHC and to foster the development of in-house expertise to sustain ongoing training and quality improvement in the provision of care for LGBT patients.
  Arms: Intervention

SUMMARY:
The primary goal of this PCORI proposal is to evaluate the impact of enhanced provider and clinical staff training to address the health disparities of SGM CHC patients to ultimately improve their health outcomes because CHCs are a key part of the U.S. health care delivery system for underserved populations. The current application proposes to test an intervention designed to understand how CHCs, including front line staff and safety net clinical providers, can identify and provide optimal care for their SGM patients, and will determine whether enhanced training of CHC staff in best practices for the provision of primary care for SGM patients will improve their clinical outcomes. The time is right for routinization of SOGI measures in EHRs and evaluation of the optimal methods to train primary care providers in the best practices for the care of SGM patients.

DETAILED DESCRIPTION:
This project will work with 12 community health centers across the country that are part of and extended from the HRSA-established Community Health Applied Research Network (CHARN) to determine the optimal way to train CHC staff in the collection of SOGI data, and will evaluate the impact of enhanced SOGI data collection on health outcomes for LGBT patients. The project will build on more than six years of collaborations of a network of safety-net CHCs, including patient investigators from the inception of the project, with a plan for ongoing local patient engagement. Aim 1: Conduct interviews with patient and clinical stakeholders regarding how SOGI data are being used to inform patient care, and how they feel SOGI data should best be collected and utilized. Aim 2: Educate providers in culturally competent patient-centered care with sexual and gender minority populations. Aim 3: Compare the effect of a SOGI educational training program to usual practice on SOGI documentation rates and appropriate screening rates for LGBT patients.

The project will determine the optimal way to train CHC staff in the collection of SOGI data, and will evaluate the impact of enhanced SOGI data collection on health outcomes for LGBT patients. The project team proposes a study design that is commonly employed to examine changes in outcomes (e.g., screening rates) across time, comparing rates prior to and after the educational training intervention. The project will measure the impact of changes to practice and to patient outcomes (e.g., depression screening, appropriate use of mammography and HPV screening for lesbians and transgender women), as well as patient satisfaction.

Results of this study would be the first of their kind to evaluate the impact of a series of educational programs on the healthcare outcomes of LGBT patients and could provide a replicable patient-centered model for routinely collecting and documenting sexual and gender minority information at CHCs and improving provider competence in care. Ultimately, the study has strong potential for improving the quality of care for sexual and gender minorities and reducing health disparities.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Clinical staff or patient at participating clinical site (for staff interviews and web surveys)
* English speakers

Exclusion Criteria:

* Does not meet the inclusion criteria above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Sexual Orientation and Gender Identity (SOGI) status | 24 month follow up period
  % of patients at CHC with SOGI status documented
Behavioral Health and Substance Use Assessment | 24 month follow up period
  Documentation of PHQ9
Behavioral Health and Substance Use Assessment | 24 month follow up period
  Documentation of AUDIT
Behavioral Health and Substance Use Assessment | 24 month follow up period
  Documentation of tobacco status
Vital Sign | 24 month follow up period
  Documentation of weight or BMI
Vaccination | 24 month follow up period
  Documentation of Hepatitis A vaccination
Vaccination | 24 month follow up period
  Documentation of Hepatitis B vaccination
Mammography | 24 month follow up period
  Documentation of mammogram
Cervical PAP | 24 month follow up period
  Documentation of PAP

SECONDARY OUTCOMES:
Behavioral health referral, if problem identified | 24 month follow up period
  Documentation of referral among those where a behavioral health problem is identified
Tobacco counselling referral, if smoker | 24 month follow up period
  Documentation of referral among current smokers
Weight control referral, if problem identified | 24 month follow up period
  Documentation of referral among those where a weight problem is identified
HIV screening | 24 month follow up period
  % of patients at CHC with HIV screening
Bacterial STI screening | 24 month follow up period
  % of patients at CHC with STI screening
Anal cancer | 24 month follow up period
  % of patients at CHC with anal PAP screening

OTHER OUTCOMES:
Patient satisfaction rates | 39 month study period
  Measured through pre- and post-intervention patient web surveys
Patient service utilization | 24 month follow up period
  Measured through annual data reports from participating sites

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Mayer, MD, Principal Investigator — Fenway Community Health Center
Locations (1):
- Fenway Community Health Cetner, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Mayer KH, Peretti M, McBurnie MA, King D, Smith NX, Crawford P, Loo S, Sigal M, Gillespie S, Davis JA, Cahill S, Grasso C, Keuroghlian AS. Training Health Center Staff in the Provision of Culturally Responsive Care for Sexual and Gender Minority Patients: Results of a Randomized Controlled Trial. LGBT Health. 2024 Feb-Mar;11(2):131-142. doi: 10.1089/lgbt.2022.0322. Epub 2023 Dec 5. PMID 38052073
- [Derived] Loo S, Peretti M, Sigal M, Noe B, Grasso C, Keuroghlian AS, Mayer KH. Health Center Leadership Perspectives Regarding Barriers to and Facilitators of Providing Culturally Responsive Care for Sexual and Gender Minority Patients. LGBT Health. 2023 Jul;10(5):391-400. doi: 10.1089/lgbt.2022.0135. Epub 2023 Feb 21. PMID 36802213
- [Derived] Mayer KH, Peretti M, McBurnie MA, King D, Smith NX, Crawford P, Loo S, Sigal M, Gillespie S, Cahill S, Keuroghlian AS, Grasso C. Wide Variability in Documentation of Sexual Orientation, Gender Identity, and Preventive Health Screenings in a Diverse Sample of U.S. Community Health Centers. LGBT Health. 2022 Nov;9(8):571-581. doi: 10.1089/lgbt.2021.0362. Epub 2022 Jun 30. PMID 35772015